CLINICAL TRIAL: NCT02827695
Title: Smart Phone Medication Adherence Saves Kidneys--SMASK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00053471
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Kidney Transplantation; Medication Adherence; Hypertension
MeSH Terms: conditions — Medication Adherence; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMASK (Experimental): Subjects will receive electronic pill tray with reminder functions activated and Bluetooth blood pressure monitor and phone app.
  Interventions: Behavioral: SMASK
- EnhancedSC (Other): Subjects will receive daily attention control texts with healthy lifestyle information and continue to use the pill tray without reminder functions.
  Interventions: Behavioral: EnhancedSC

INTERVENTIONS:
Behavioral: SMASK — Medication adherence and BP monitoring
  Arms: SMASK
Behavioral: EnhancedSC — Standard care without med reminder functions with healthy lifestyle texts
  Arms: EnhancedSC

SUMMARY:
Investigators will employ a 2-arm Randomized Controlled Trial (RCT) design with the subject as the unit of randomization and analysis. Kidney transplant recipients having uncontrolled hypertension will be enrolled into a screening phase to measure medication non-adherence. Each subject will use an electronic pill tray for 1 month without any reminder functions activated. Non-adherent subjects who remain uncontrolled will be randomly assigned to SMASK or Standard Care (SC). SC will continue to use the pill tray with reminders turned off and will receive attention control texts with healthy lifestyle information. SMASK will have the reminder functions of the electronic pill tray activated and will receive a Bluetooth blood pressure monitor and an app to collect the data and send to researchers.

Subjects in the second phase will participate in 4 more evaluations at months 1, 3, 6, 12 post randomization. Research staff will measure resting blood pressure and heart rate.

DETAILED DESCRIPTION:
A randomized RCT will be conducted with kidney transplant patients identified as hypertensive (>129 SBP following KDIGO guidelines) via medical history. Those identified as being nonadherent for 4 weeks during the first month post enrollment (adherence score <0.85) will be eligible to participate in the second phase. Participants in the second phase will be randomly assigned to standard care (SC) + attention control or the mHealth program plus SC.

Following informed written consent, eligible patients will be asked to complete several brief surveys aimed at determining, mood state, perceived stress, self-efficacy assessment, comfort with mHealth devices, perceptions of treatment burden and attitudes towards mhealth. Subjects will have their blood pressure measured and if SBP is >129 they will enter the screening phase. Subjects will be provided a Medication dispensing device system. Subjects will be called the following day to check if there were any problems in filling the Simplemed tray.

The Simplemed has four compartments for each day of the week for potential use. Microelectronic circuitry in each compartment on the tray date stamps the opening of each compartment and removal of the refill tray. These signals are relayed via an internal modem to a server for processing. Data can then be sent directly into the MUSC server that compiles individuals' health data from multiple delivery points. Adherence rate across the first month will be calculated at weekly intervals.

All subjects will return for a visit at the end of their 4 week screening period. Those with an adherence score <0.85 for 4 weeks and whose SBP continues to be >129 will be invited to participate in the second phase of the RCT. Evaluations performed at this visit will include anthropometrics, questionnaires, and resting BP. A Spacelabs ABP monitor will be applied with instructions for wearing the monitor 24 hrs. The subjects will be randomized to SMASK+SC or SC+ attention control groups after the baseline procedures are completed. Those with med adherence score ≥0.85 or who have SBP ≤ 129 will return their pill tray but not proceed into the second phase. Recruitment will end when 80 subjects have successfully transitioned into the second phase (RCT) of the study.

The SC+ attention control group will continue to use Simplemed with reminder functions disabled, they will be sent daily text messages or links to PDF documents or videos containing health information as attention control. The SMASK mhealth intervention group will also receive SC and have the Simplemed reminder functions turned on (blink for ½ hr when medication is due, chime additional ½ hr, then text or email after 1 hour) and receive training in use of the A&D BP monitor. They will be instructed to measure their blood pressure twice daily AM, PM) on at least every third day. Patients will be provided with and shown how to use the smart phone app and activate the app when they record their blood pressure readings.

ELIGIBILITY:
Inclusion Criteria:

1. ≥21 years old;
2. First time recipient of a functioning solitary kidney transplant;
3. Prescribed ≥3 medications for immunosuppression and HTN;
4. Transplant MD's assent that patient is able to participate;
5. Ability to speak, hear and understand English;
6. Able to take their own BP;
7. Self-administers medications;
8. SBP >129 mmHg at clinic visit(s) in 4 weeks prior, and at initial study evaluation at enrollment;
9. ***Only subjects with adherence score <.85 after 1-month screening and SBP >129 mmHg at baseline will be randomized.

Exclusion Criteria:

1. Failure to meet any inclusion criterion;
2. Ongoing substance abuse (e.g., >21 alcoholic drinks/week);
3. Psychiatric illness requiring treatment beyond antidepressants;
4. Will attempt to become pregnant within the year;
5. Pregnant or nursing women, prisoners, and institutionalized persons.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05; Primary Completion 2020-05 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | six months
  % with electronic monitor-derived adherence scores >.90;

SECONDARY OUTCOMES:
Provider adherence to KDIGO guidelines | six months
  measured by timing of medication changes
Changes in Self-Determination Theory mediators | six months
  Survey responses demonstrate increased (e.g., perceived competence and autonomous regulation).
BP control | Six months
  % reaching and sustaining Kidney Disease Improving Global Outcomes (KDIGO) guidelines for BP control (resting and 24-hr BP<130/80 mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: John McGillicuddy, MD, Principal Investigator — MUSC Transplant Surgery
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829